CLINICAL TRIAL: NCT06520332
Title: Comparative Evaluation of the Clinical Efficacy of Short Implants With Standard-Length Implants Placed in Native/Augmented Bone of the Patients With a History of Periodontitis - A Randomised Controlled Trial
Brief Title: Comparative Evaluation of the Clinical Efficacy of Short Implants With Standard-Length Implants - a Randomised Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02_D012_00040
Record Dates: First submitted 2024-07-19; First posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Dental Implant
Keywords: Dental implant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 10 Short implants will be placed in the residual vertical bone height of 5 to 8mm . (Experimental): One short dental implant will be placed whose length will be less than or equal to 6mm.
  Interventions: Procedure: Dental Implant Surgery - short implant group (less than or equal to 6mm)
- 10 Standard implants of length ≥ 10mm will be placed in augmented/native bone . (Active Comparator): This Conventional Dental implant group will act as control.
  Interventions: Procedure: Dental Implant Surgery - Conventional implant group (greater than or equal to 10mm)

INTERVENTIONS:
Procedure: Dental Implant Surgery - short implant group (less than or equal to 6mm) — A mucoperiosteal flap will be raised in edentulous ridge. A short dental implant (experimental group) will be placed according to the standard protocol.
  The platform of the implant will be placed 2 to 3 mm below CEJ of adjacent teeth.
  The surgical wound closure will be coapted with mattress and single interrupted sutures
  Arms: 10 Short implants will be placed in the residual vertical bone height of 5 to 8mm .
Procedure: Dental Implant Surgery - Conventional implant group (greater than or equal to 10mm) — A mucoperiosteal flap will be raised in edentulous ridge. A standard length implant ( comparative group) ( ≥10mm) will be placed according to the standard protocol in the augmented/native bone .
  The platform of the implant will be placed 2 to 3 mm below CEJ of adjacent teeth.
  The surgical wound closure will be coapted with mattress and single interrupted sutures
  Arms: 10 Standard implants of length ≥ 10mm will be placed in augmented/native bone .

SUMMARY:
Periodontal disease , especially in its advanced stages , is one of the main cause for tooth loss .Tooth replacement options include dental implants , fixed partial denture , removable partial denture and complete dentures . Dental implants have become more common treatment for replacing missing teeth and aim to improve chewing efficiency, physical health and esthetic. Although conventional implants cannot be placed in every site due to resorption of the alveolar socket after extraction. Thus short implants can be used as an alternative . Hence, this study aims at comparing the clinical efficacy of short implants with standard length implants placed in native or augmented bone in patients with a history of periodontitis.

DETAILED DESCRIPTION:
Implant supported prosthesis have proven as an esthetic , functional restoration with long term predictability by re-establishing appearance , comfort and mastication .

Following extraction , the bony socket undergoes significant horizontal and vertical reduction . This 3D resorption of alveolar sockets after extraction often lead to limitations for implant placement . Severe ridge atrophy complicates rehabilitation of posterior edentulous regions . This lack of adequate bone necessitates additional reconstructive surgeries such as guided bone regeneration, vertical ridge augmentation , sinus floor elevation , block grafts , distraction osteogenesis and transposition procedures of the inferior alveolar nerve to allow anatomically sound placement of dental implants . These complex surgical procedures can result in intra-operative complications like infections of graft/membranes and it's exposure and post-operative complications such as swelling , pain , nerve disturbances with an associated increased reluctance of the patient to undergo them . Also these procedures, has significantly increased treatment duration, morbidity, risk of complications and costs.

Currently , alternative procedures to avoid these additional surgeries and the associated complications encourages the use of less invasive procedures such as short implants. Short implant placements can reduce morbidity and recovery time associated with bone augmentation procedures. Thus use of shorter dental implant has shown to be a plausible solution in cases of confined space , as well as those associated with unavoidable anatomical structures , such as lingual concavities or the maxillary sinus proximation which can be prone to surgical difficulties. Short implants offer a minimally invasive approach with ease of handling , reduced surgical invasiveness and low risk of trauma to vital structures . Evidence suggests that short implants could decrease implant failure , marginal bone loss , biological complications and improve patient satisfaction. The evidence from the literature must be interpreted with caution due to the variable protocols. Clinicians require a thorough comprehension of implant dentistry to achieve predictability.Thus there is a need for well designed RCT's analysing and comparing the clinical outcomes of short implants placed in native bone with long implants placed in native or augmented bone .

Thus, the aim of the current randomised controlled clinical trial (RCT) study will be to analyse the clinical efficacy of short implants (≤6 mm) and compare it with standard length implants (≥10mm) placed in native / augmented bone in patients with history of periodontitis.

ELIGIBILITY:
Inclusion Criteria:

1. Age group - 18 years and above
2. Presence of >2 mm keratinised tissue to allow flap management.
3. Systemically healthy patients
4. The residual vertical bone height at the implant sites ranging from 6 to 9 mm for short implant placement ; > 9 mm for standard implant placement.
5. History of periodontitis

Exclusion Criteria:

1. Medical conditions contraindicating surgical interventions

   1. Uncontrolled diabetes
   2. Hemorrhagic disorders
2. Intravenous and oral bisphosphonate therapy.
3. Irradiation in head and neck
4. Pregnant and lactating women
5. Subjects with known bone metabolic disorders (paget's disease , fibrous dysplasia etc.)
6. Known smokers and alcoholics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
The primary outcome that will be assessed is implant survival rate. | 6 months
  The primary objective of this randomised controlled clinical trial will be to compare the survival rate of short implants (≤ 6 mm ) and standard-length implants (≥ 10 mm) in patients with a history of periodontitis; through clinical and radiographic analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Krishnadevaraya college of dental sciences, Bangalore, Karantaka, India

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared with other researchers.

REFERENCES:
- [Background] Esposito M, Barausse C, Pistilli R, Sammartino G, Grandi G, Felice P. Short implants versus bone augmentation for placing longer implants in atrophic maxillae: One-year post-loading results of a pilot randomised controlled trial. Eur J Oral Implantol. 2015 Autumn;8(3):257-68. PMID 26355170